CLINICAL TRIAL: NCT02926105
Title: Comparison of the Effects of Three Home-based Exercise Programmes Regarding Falls, Quality of Life and Exercise-adherence in Older Adults at Risk of Falling: Protocol for a Randomised Controlled Trial
Brief Title: Comparison of Home-based Exercise Programmes for Falls Prevention and Quality of Life in Older Adults
Acronym: SwissCHEF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: Fondation Leenaards, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-00931
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Accidental Falls

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T&E Home-based exercise programme (Experimental): Individually tailored home-based test and exercise programme
  Interventions: Behavioral: T&E Home-based exercise programme
- Otago (Experimental): Individually tailored exercise programme
  Interventions: Behavioral: Otago
- Helsana booklet (Active Comparator): Helsana recommendations and exercises
  Interventions: Behavioral: Helsana booklet

INTERVENTIONS:
Behavioral: T&E Home-based exercise programme — "T&E" exercises programme consists of home-based individually tailored balance and functional strength tests and exercises performed 3x a week over 12 months, accompanied by eight in-home visits of physiotherapists during the first six months.
  Other Names: T&E
  Arms: T&E Home-based exercise programme
Behavioral: Otago — Otago exercises programme consists of home-based individually tailored balance, strength and walking exercises performed 3x a week over 12 months, accompanied by eight in-home visits of physiotherapists during the first six months.
  Arms: Otago
Behavioral: Helsana booklet — Helsana programme consists of a booklet with recommendations and 10 exercises performed 3x a week over 12 months.
  Other Names: Helsana
  Arms: Helsana booklet

SUMMARY:
This study compares the effects of three home-based exercise programmes in "at-risk to falling" older adults living in their own home on the incidence of falls (number and severity), risk factors, and quality of life as well as on the adherence to exercise. The subjects will be randomized and allocated in three groups. The group A will receive the "Test-and-Exercise" home-based programme (T&E), the group B will receive the "Otago" home-based exercise programme and the group C (activ-control group) will receive the "Helsana" booklet

DETAILED DESCRIPTION:
Home-based exercise programmes appear to reduce rate of falls, number of fallers, risk of falling and risk of death and to improve balance, leg strength, function, physical activity and balance confidence in older adults living in the community.

The Test-and-Exercise home-based programme (T&E) contains 50 tests and 50 exercises to improve balance, strength and ability in older adults. It is especially built for older adults and is based on the concept of self-efficacy and empowerment. The originality of this programme is the evaluation of the difficulty perceived of the balance-exercises. It is delivered on a booklet which investigators had good experience with in our pilot study, with pictures and descriptions of each test and each exercise. Investigators also developed a mobile application. This application will be transmitted on a tablet-computer. In addition, the participants will receive cards with pictures of the exercises, to put into a plastic sheet to have an overview of their own exercise programme. This programme will be implemented from especially trained physiotherapists.

The Otago home-based exercise programme was developed in New-Zeeland in the 2000's to prevent falls in older adults. It proposes 22 exercises and walk training. The physiotherapists give an exercise prescription at each home visit. It shows good results for decrease falls in older adults, but the exercise adherence decrease also with the time.

The Otago home-based exercise programme was developed in New-Zeeland in the 2000's to prevent falls in older adults. It proposes 22 exercises and walk training. The physiotherapists give an exercise prescription at each home visit. It shows good results for decrease falls in older adults, but the exercise adherence decrease also with the time.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and older,
* Living in their own home,
* Having a history of fall in the previous 12 months or perceiving fear of falling (≥ 20 points on FES-I,
* Being able to walk without auxiliary tools in their home.
* Signed Informed Consent

Exclusion Criteria:

* Having severe vision impairment that do not permit the reading of the exercise-programme booklet and that do not permit the completing of the monthly diaries,
* Receiving physiotherapeutic treatment with balance learning,
* Having cognitive impairment (<25 points on the Mini-Mental State Examination (MMSE) of Folstein

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
number of falls | one year

SECONDARY OUTCOMES:
Fear of falling | one year
  FES-I
Severity of falls | one year
  Scale of Schwenk 2012
Risk of fall | one year
  Algorithm STEADI
Quality of life | one year
  OPQOL-35
Exercise adherence | one year
  Monthly calender

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gabrielle Mittaz Hager, MS, Principal Investigator — HES-SO Valais-Wallis
Locations (3):
- Switzerland (3):
  - CUTR Sylvana, Épalinges, Canton of Vaud
  - Physiotherapie Nevzati, Zurich, Canton of Zurich
  - HES-SO Valais-Wallis, Leukerbad, Valais

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hager AM, Mathieu N, Carrard S, Bridel A, Wapp C, Hilfiker R. Partially supervised exercise programmes for fall prevention improve physical performance of older people at risk of falling: a three-armed multi-centre randomised controlled trial. BMC Geriatr. 2024 Apr 3;24(1):311. doi: 10.1186/s12877-024-04927-0. PMID 38570773
- [Derived] Mittaz Hager AG, Mathieu N, Lenoble-Hoskovec C, Swanenburg J, de Bie R, Hilfiker R. Effects of three home-based exercise programmes regarding falls, quality of life and exercise-adherence in older adults at risk of falling: protocol for a randomized controlled trial. BMC Geriatr. 2019 Jan 14;19(1):13. doi: 10.1186/s12877-018-1021-y. PMID 30642252
- See also: Trial homepage — http://www.swiss-chef-trial.ch